CLINICAL TRIAL: NCT00178191
Title: A Randomized Trial of Botox for Severe Urge Incontinence
Brief Title: Randomized Trial for Botox Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michael Flynn, MD, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10466; 1R21AG025490-01 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Surveys and Questionnaires; Urodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 200 units Botox (Experimental): 200 units Botulinum-A toxin
  Interventions: Other: Bladder diary; Other: Questionnaires; Procedure: Urodynamics; Other: Pad weight
- 300 units Botox (Experimental): 300 units Botulinum-A toxin
  Interventions: Other: Bladder diary; Other: Questionnaires; Procedure: Urodynamics; Other: Pad weight
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Bladder diary; Other: Questionnaires; Procedure: Urodynamics; Other: Pad weight

INTERVENTIONS:
Other: Bladder diary — 3-day bladder diary
Other: Questionnaires — Incontinence Quality of Life questionnaires
Procedure: Urodynamics — Urodynamics
Other: Pad weight — Pad weight

SUMMARY:
The purpose of this study is to determine how effective Botox is in reducing the amount of urine leaked and which dose of Botox is more effective and safe in those who have urinary urge incontinence.

DETAILED DESCRIPTION:
The prevalence of urinary incontinence in the US ranges from 3-14% with epidemiologic estimates ranging widely.1 Most urinary incontinence can be categorized into stress urinary incontinence (SUI) or UUI with UUI remaining more common and debilitating than SUI.2 A major cause of UUI is overactive bladder or detrusor instability (DI), and while DI is very common, its etiology remains unknown. DI is often successfully managed with behavioral therapy, physical therapy, medications and surgery with the most effective therapy being anticholinergic medication.2 However, side effects including dry mouth, and constipation often lead to discontinuation of these drugs. In addition, many patients fail anticholinergic medication and have persistent urinary leakage. Women who fail these treatments have limited options.

ELIGIBILITY:
Inclusion Criteria: Subjects must have ALL of the following:

* Completed a routine evaluation of incontinence (urodynamics, bladder diaries, and pad weights) through the urogynecology clinic at SMH within 3 months of the screening visit
* Symptoms of urge incontinence associated with leakage on bladder diary
* 24-hour pad weight >100 cc's (volume requiring multiple daily diaper changes)
* Absence of a bladder infection or other condition that could explain urinary leakage
* Absence of stress incontinence or a cough leak point pressure > 100 cm H2O on cystometry (this correlates with mild stress incontinence)
* Failed anticholinergic therapy
* Willingness and ability to perform intermittent clean catheterization (due to the risk of prolonged urinary retention from Botox)
* The ability and willingness to return for surveillance evaluations
* A negative urine pregnancy test if at risk for pregnancy
* Competent to give signed consent and complete all of the study measures

Exclusion Criteria:

* Children (< 21 years old), pregnant women and prisoners
* History of carcinoma of the bladder
* Absence of a measurable detrusor contraction on a pressure flow micturition study
* A foreign body in the bladder or other correctable etiology for the UUI
* Prior documented resistance to Botox
* Gross fecal incontinence (due to confounding effects on pad weights and counts)
* Known allergy to lidocaine or related compounds (used for local analgesia)
* Known allergy to or inability to take both Bactrim DS or Ciprofloxacin (used for urinary tract infection prophylaxis)
* Current use of an aminoglycoside or preparing for general anesthesia within 1 week (risk of synergetic effects
* Known neurologic conditions such as Parkinson's disease, myasthenia gravis, multiple sclerosis, autonomic dysfunction, Lambert-Eaton syndrome, Amyotrophic Lateral Sclerosis or other neurologic disorder that may impact urinary function or the effect of Botox.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Flynn, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started June, 2005 and completed Dec, 2007
Period: Overall Study
Arm/Group | 200 Units Botox | 300 Units Botox | Placebo
Started | 11 | 10 | 7
Completed | 11 | 10 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 Units Botox | 300 Units Botox | Placebo | Total
Number analyzed (Participants) | 10 | 11 | 7 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0.0
  Between 18 and 65 years | 2 | 8 | 2 | 12.0
  >=65 years | 8 | 3 | 5 | 16.0
Age Continuous [Mean (Standard Deviation); unit: years] | 76.20 (10.65) | 61.72 (13) | 74.14 (11.01) | 70 (13.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 7 | 28.0
  Male | 0 | 0 | 0 | 0.0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 7 | 28.0

OUTCOME MEASURES:

1. Primary Outcome: Episodes/Day
Description: number of incontinence episodes/day
Time Frame: 9 months
Measure: Mean (Standard Error); unit: number
Arm/Group | 200 Units Botox | 300 Units Botox | Placebo
Number analyzed (Participants) | 11 | 10 | 7
number | 6.6 (0.9687) | 3.52 (0.95) | 8.7 (1.52)

ADVERSE EVENTS:
Arm/Group | 200 Units Botox | 300 Units Botox | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/7

LIMITATIONS AND CAVEATS:
Please see published manuscripts for additional details

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No